CLINICAL TRIAL: NCT06026358
Title: Tirbanibulin 1% Ointment for the Treatment of Actinic Keratosis on the Back of the Hands. An Internally Placebo Controlled, Partly Blinded Clinical Pilot Study
Brief Title: Tirbanibulin 1% Ointment for the Treatment of Actinic Keratosis on the Back of the Hands
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of ressources
Sponsor: Medical University of Graz (Other)
Collaborators: Almirall, SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tirbanibulin: Back of Hands
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — tirbanibulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirbanibulin (Experimental): Treatment
  Interventions: Drug: Tirbanibulin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Tirbanibulin

INTERVENTIONS:
Drug: Tirbanibulin — subjects receive 2,5 mgTirbanibulin in 250 mg ointment with daily administration of one single sachet on the left hand and 250mg ointment placebo on the right hand for 5 d in a single-blinded manner.

SUMMARY:
Interventional, monocentric, national, internal placebo-controlled, prospective pilot study, consisting of two parts, A (single-blinded) and B (open) to assess Efficacy of Tirbanibulin for the treatment of AK on the back of the hand. In part A, eligible subjects receive Tirbanibulin on the left hand and placebo on the right hand for 5 d in a single-blinded manner. Safety and efficacy are assessed at day 8 (± 1 d) (3 days after the end of treatment (EoT+3) and day 57 (± 7 d) after the start of the treatment. Pictures will be taken at baseline, 8 d and 57 d (± 7 d) as per protocol and optional during unscheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* o Informed consent

  * Diagnosed with AK on both hands
  * 4-8 AK lesions on each hand, difference in number of lesions < 20%
  * Grade of lesions comparable in both hands: non hypertrophic, non-hyperkeratotic
  * Willing and able to comply with all study procedures
  * Use of medically acceptable contraception (both sexes)
  * 18 - 99 years of age.

Exclusion Criteria:

* o History of sensitivity and/or allergy to any of the ingredients in the study medication.

  * Open lesions of any kind on the hands
  * Concomitant cutaneous malignancy in treatment area
  * Immune deficiency
  * Participation in another clinical trial during the last 6 months
  * Had been previously treated with Tirbanibulin
  * Anticipated need for in-patient hospitalisation or in-patient surgery from Day 1 to Day 57.
  * Treatment with 5-fluorouracil (5-FU), imiquimod, diclofenac, photodynamic therapy, or other treatments for AK within the treatment area or within 2 cm of the treatment area within 8 weeks prior to the Screening Visit.
  * Use of the following therapies and/or medications within 2 weeks prior to the Screening Visit:

    * Cosmetic or therapeutic procedures (eg, use of liquid nitro-gen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within the treatment area or within 2 cm of the selected treat-ment area
    * Acid-containing therapeutic products (eg, salicylic acid or fruit acids, such as alpha and beta-hydroxyl acids and gly-colic acids), topical retinoids, or light chemical peels within the treatment area or within 2 cm of the selected treat-ment area
    * Topical salves (nonmedicated/nonirritant lotion and cream were acceptable) or topical steroids within the treatment area or within 2 cm of the selected treatment area; artifi-cial tanners within the treatment area or within 5 cm of the selected treatment area.
  * Use of the following therapies and/or medications within 4 weeks prior to the Screening Visit:

    * Treatment with immunomodulators (eg, azathioprine), cy-totoxic drugs (e.g., cyclophosphamide, vinblastine, chlo-rambucil, methotrexate) or interferons/interferon induc-ers.
    * Treatment with systemic medications that suppress the im-mune system (e.g., cyclosporine, prednisone, methotrex-ate, alefacept, infliximab).
  * Use of systemic retinoids (e.g., isotretinoin, acitretin, bexaro-tene) within 6 months prior to the Screening Visit.
  * Skin disease (e.g., atopic dermatitis, psoriasis, eczema) or con-dition (e.g., scarring, open wounds) that, in the opinion of the investigator, might interfere with the study conduct or evalu-ations, or which exposed the subject to unacceptable risk by study participation.
  * Other significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the Investigator, would have exposed the subject to unacceptable risk by study participa-tion.
  * Pregnancy or lactation
  * Excessive exposure to UV radiation during study period.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Partial clearance at day 57 ± 7 after start of blinded treatment | day 57 ± 7 after start of blinded treatment

IPD SHARING:
Plan to Share IPD: No